CLINICAL TRIAL: NCT06838156
Title: Comparison of Analgesic Efficacy of Quadratus Lumborum Type 3 and Suprainguinal Fascia Iliaca Compartment Block in Total Hip Arthroplasty Surgery: a Randomized Controlled Trial
Brief Title: Comparison of Analgesic Efficacy of Quadratus Lumborum Type 3 and Suprainguinal Fascia Iliaca Compartment Block in Total Hip Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Muzaffer GENCER, Associate Professor Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GK-QLB-SIFI
Record Dates: First submitted 2025-02-09; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Opioid Consumption; Pain Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIFI Group (Active Comparator): Group of 30 patients who underwent SIFI block
  Interventions: Drug: Bupivacain
- QLB Type 3 (Active Comparator): Group of 30 patients who underwent QLB block
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — Suprainguinal Fascia Iliaca Compartment block was performed with a linear probe placed over the inguinal ligament using a portable ultrasound device. After visualization of the femoral nerve, 30 ml of 0.25% bupivacaine was injected into the fascia iliaca overlying the iliopsoas muscle using an appropriate needle.
  Other Names: SIFI
  Arms: SIFI Group
Drug: Bupivacain — Quadratus Lumborum Type 3 block was performed using a portable ultrasound device with a linear probe placed between the costal margin and the iliac crest on the lateral abdominal wall. 30 ml of 0.25% bupivacaine was injected between the quadratus lumborum and psoas muscles using an appropriate needle.
  Other Names: QLB Type 3
  Arms: QLB Type 3

SUMMARY:
Total Hip Arthroplasty (THA) is a complex surgical procedure frequently performed to treat degenerative conditions in the hip joint. As people's life expectancy increases, the need for hip arthroplasty increases. İnvestigetors aimed to compare the analgesic properties of SIFI and QLB blocks.

ELIGIBILITY:
Inclusion Criteria:

1. Elective patients scheduled for hip arthroplasty surgery
2. Patient willingness to participate in the study
3. Patients over 18 years age of, ASA I-II-III,

Exclusion Criteria:

1. Patients not wanting to participate in the study
2. Patients who do not want regional anesthesia technique
3. Allergic or coagulated patients
4. Patients with liver, kidney, lung, heart failure and septic patients
5. Neurological disorder, history of convulsions
6. ASA IV patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Effect on pain score | At 1,2,4, 6, 12 and 24 hours after surgery
  Postoperative 24-hour Visual Analog Scale was measured. ( 0=best 10=worst)

SECONDARY OUTCOMES:
Opioid Consumption | At 1,2,4, 6, 12 and 24 hours after surgery
  Intravenous patient-controlled analgesia (PCA) with tramadol was administered to both groups in the postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam Ve Sakura City Hospital, Başakşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Safa B, Trinh H, Lansdown A, McHardy PG, Gollish J, Kiss A, Kaustov L, Choi S. Ultrasound-guided suprainguinal fascia iliaca compartment block and early postoperative analgesia after total hip arthroplasty: a randomised controlled trial. Br J Anaesth. 2024 Jul;133(1):146-151. doi: 10.1016/j.bja.2024.04.019. Epub 2024 May 18. PMID 38762396
- [Background] Xia Q, Ding W, Lin C, Xia J, Xu Y, Jia M. Postoperative pain treatment with transmuscular quadratus lumborum block and fascia iliaca compartment block in patients undergoing total hip arthroplasty: a randomized controlled trial. BMC Anesthesiol. 2021 Jul 10;21(1):188. doi: 10.1186/s12871-021-01413-7. PMID 34243719